CLINICAL TRIAL: NCT02786446
Title: Comparison of Different Analgesia Drug Regimens for Pain Control During ESWL for Renal Stones: A Randomized Control Study
Brief Title: Comparison of Different Analgesia Drug Regimens for Pain Control During ESWL for Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Waqas, Post Graduate Trainee, Shifa International Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ShifaIH
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Renal Stone
Keywords: Lidocaine gel; Extracorporeal shockwave lithotripsy; Naproxen sodium; Pain score
MeSH Terms: conditions — Nephrolithiasis | interventions — Naproxen; Anti-Inflammatory Agents, Non-Steroidal; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lidocaine gel (Active Comparator): 20 grams Lidocaine gel 2 % will be applied to corresponding lumber area of the patients 30 minutes before undergoing ESWL for renal stone.Max 4000 shockwaves will be administered. Rescue intravenous nalbuphine will be administered during procedure.Visual analogue pain score will be measured after completion of procedure or during procedure just before giving rescue iv analgesia if needed.
  Interventions: Drug: Lidocaine gel,
- Naproxen Sodium (Active Comparator): Oral Naproxen sodium 550 mg will given to patients 45 minutes before ESWL for renal stones.Max 4000 shockwaves will be administered. Rescue intravenous nalbuphine will be administered during procedure.Visual analogue pain score will be measured after completion of procedure or during procedure just before giving rescue iv analgesia if needed.
  Interventions: Drug: Naproxen Sodium
- Lidocaine Gel and Naproxen Sodium (Active Comparator): Oral Naproxen sodium 55o mg and locally applied 2 % lidocaine gel to patients before ESWL for renal stones.Max 4000 shockwaves will be administered. Rescue intravenous nalbuphine will be administered during procedure.Visual analogue pain score will be measured after completion of procedure or during procedure just before giving rescue iv analgesia if needed.
  Interventions: Drug: Lidocaine gel and Naproxen Sodium

INTERVENTIONS:
Drug: Lidocaine gel, — 2% lidocain gel will be applied to coresponding lumber area 30 minutes before ESWL for renal stones. Maximum of 4000 shock waves will be delivered. Rescue analgesia will be given as intravenous nalbuphine if patient demanded. Pain score is measured with visual analogue pain score from 1 to 10 after completion of procedure if patient donot needed rescue analgesia and during procedure just before giving rescue analgesia in those who demanded it.
  Other Names: Lignicaine
  Arms: Lidocaine gel
Drug: Naproxen Sodium — Tab Naproxen sadium 550 mg per oral will be given to patients 30 minutes before ESWL for renal stones. Maximum of 4000 shock waves will be delivered. Rescue analgesia will be given as intravenous nalbuphine if patient demanded. Pain score is measured with visual analogue pain score from 1 to 10 after completion of procedure if patient donot needed rescue analgesia and during procedure just before giving rescue analgesia in those who demanded it.
  Other Names: NSAIDS
  Arms: Naproxen Sodium
Drug: Lidocaine gel and Naproxen Sodium — Tab Naproxen sodium 550 mg per oral will be given to patients 45 minutes before ESWL and 2% lidocain gel will be applied to coresponding lumber area 30 minutes before ESWL for renal stones. Maximum of 4000 shock waves will be delivered. Rescue analgesia will be given as intravenous nalbuphine if patient demanded. Pain score is measured with visual analogue pain score from 1 to 10 after completion of procedure if patient donot needed rescue analgesia and during procedure just before giving rescue analgesia in those who demanded it.
  Other Names: NSAIDS and Lidocaine
  Arms: Lidocaine Gel and Naproxen Sodium

SUMMARY:
We want to compare the effect of lignocaine 2 % gel, Naproxen sodium and their combination on the pain control during extracorporial shock wave lithotripsy for renal stones.

DETAILED DESCRIPTION:
Introduction of ESWL (extracorporeal shock wave lithotripsy) has revolutionized the treatment of urolithiasis due to its noninvasive in nature, cost effectiveness, reduced hospitalization time and less morbidity1, 2.Impact of shock waves cause pain in most of the patient requiring analgesia or sedation. It is important to make patient pain free to get the maximum possible stone free rates3, 4. Opioids are used most commonly for pain relief in ESWL but with side effects requiring patient monitoring and delayed hospital stay3, 4. NSAIDS also showed promising results regarding pain control in ESWL without side effects of opoids1, 5. Local analgesia gels have controversial role in relieving pain in ESWL 1, 6. There are yet no guidelines for pain relief during ESWL1, 4. We intend to compare the effect of local analgesia gel, oral NSAIDS and their combination on pain during lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years Having renal stone Meet the criteria for ESWL

Exclusion Criteria:

* H/o chronic use of analgesia, 2) Allergy to any of the used medications, 3) those having ureteric stones, 4) Serum creatinine>1.4, 5) Pregnant patients, 6) having gastric ulcer disease, 7) not willing to participate, 8) Have coagulopathy and 9) active urinary-tract infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean pain score | During or immediately after procedure
  Pain score will be assessed immediately after completion of ESWL for those who will not need rescure intravenous analgesia and immediately just beforegiving rescue analgesia in those who needed it.

IPD SHARING:
Plan to Share IPD: No